CLINICAL TRIAL: NCT03703037
Title: Clinical Utility of Uterine, Fetal Cerebral Doppler and Oligohydramnios to Predict Abnormal Heart Rate Tracings in Pregnancies at or Beyond 41 Weeks
Brief Title: Uterine, Fetal Cerebral Doppler and Oligohydramnios to Predict Abnormal Heart Rate Tracings in Postterm Pregnancies
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Flavio Hernández Castro, Principal investigator Flavio Hernández Castro MD PhD, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: GI17-00009
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Abnormality in Fetal Heart Rate or Rhythm; Ultrasound; Late Pregnancy
Keywords: Late term pregnancy; Doppler
MeSH Terms: interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort: This will be a nested case-control study. Women with low risk pregnancies at or beyond 41 weeks, who will be referred to our Maternal-fetal unit and admitted 1 to 2 days prior to induction of labour according institutional protocol will constitute the cohort.
  Then women with intrapartum abnormal fetal heart rate tracings (cases) will be identified and match with controls. The primary outcome will be to obtain odds ratios for the Doppler ultrasound parameters (middle cerebral artery pulsatility index, mean uterine artery pulsatility index and Middle cerebral artery pulsatility index to mean uterine artery pulsatility index ratio) and Ultrasound assessment of amniotic fluid index that would be associated with intrapartum category III fetal heart rate tracing.
  Interventions: Diagnostic Test: Ultrasound and Doppler ultrasound
- Cases: Cases will be patients with abnormal intrapartum cardiotocogram (category III fetal heart rate tracing).
  Intervention: Ultrasound and Doppler ultrasound
  Interventions: Diagnostic Test: Ultrasound and Doppler ultrasound
- Controls: Those will be patients with normal intrapartum cardiotocogram (category I fetal heart rate tracing) or category II that converted into category I after intrauterine resuscitation methods.
  Intervention: Ultrasound and Doppler ultrasound
  Interventions: Diagnostic Test: Ultrasound and Doppler ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound and Doppler ultrasound — Assessment of fetal cerebral and maternal uterine pulsatility index using Doppler ultrasound. Measurement of amniotic fluid index according to four-quadrant technique.
  Other Names: Pulsatility index; Amniotic fluid index

SUMMARY:
Objective: To estimate the value of uterine, fetal cerebral Doppler and oligohydramnios to predict abnormal fetal heart rate tracings in pregnancies at or beyond 41 weeks

DETAILED DESCRIPTION:
This will be a nested case-control study that was conducted at University Hospital Dr. Jose E. Gonzalez after the approval of Institutional ethical committee. Women with low risk late term or postterm pregnancy (at least 41 weeks) with confirm gestational age who will be referred to our Maternal-fetal unit and admitted 1 to 2 days prior to induction of labour according institutional protocol will be recruited and constitute the cohort.

Cases will be patients with abnormal intrapartum cardiotocogram (category III fetal heart rate tracing). For each case, four controls will be matched. The primary outcome will be to obtain odds ratios for the Doppler parameters (middle cerebral artery pulsatility index, mean uterine artery pulsatility index and Middle cerebral artery pulsatility index to mean uterine artery pulsatility index ratio) and amniotic fluid index that would be associated with intrapartum category III fetal heart rate tracing.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age of at least 287 days (41 weeks)
* Low risk pregnancy (defined as the absence of maternal or fetal complications other than postterm pregnancy)

Exclusion Criteria:

* Twin or multiple gestation
* Uncertain gestational age
* Non vertex presentation
* Estimated fetal weight below the 10th percentile for gestational age (Hadlock´s formula)
* Fetal macrosomia (estimated fetal weight ≥ 4 Kilos) diagnosed by clinical measurement (Johnson´s technique) or ultrasound measurement (Hadlock´s formula).
* Fetal abnormalities found on routine anomaly scan.
* Maternal medical disorder (preeclampsia, chronic hypertension, diabetes, lupus, hyperthyroidism)
* Prelabour rupture of membranes
* Antepartum hemorrhage
* Any fetopelvic disproportion that could create dystocia during labor.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with low risk late term or postterm pregnancy (at least 41 weeks) with confirm gestational age by first trimester ultrasound examination, who will be referred to our Maternal-fetal unit and admitted 1 to 2 days prior to induction of labour according institutional protocol.
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Category III fetal heart rate tracings | 24 hours
  Absent baseline fetal heart rate variability and any of the following: recurrent late decelerations, recurrent variable decelerations, bradycardia, sinusoidal pattern

SECONDARY OUTCOMES:
Middle cerebral artery pulsatility index | 24 hours before delivery
  The middle cerebral artery pulsatility index will be obtained in a transversal view of the fetal head, at the level of its origin from the circle of Willis. Measurements will be obtained during periods of fetal apnea, and the angle of insonation will be maintained as close to 0° as possible when interrogating the middle cerebral artery
Mean uterine artery pulsatility index | 24 hours before delivery
  The probe will be placed on the lower quadrant of the abdomen, angled medially, and again color Doppler imaging will be used to identify the uterine artery at the apparent crossover with the external iliac artery. Measurements will be taken approximately 1 cm distal to the crossover point. In all cases, once it had been ensured that the angle was less than 20◦, the pulsed Doppler gate will be placed over the whole width of the vessel. Angle correction was then applied and the signal updated until three to five similar consecutive waveforms had been obtained. Mean pulsatility index will be calculated as the average pulsatility index of right and left arteries.
Middle cerebral artery pulsatility index to mean uterine artery pulsatility index ratio | 24 hours before delivery
  The ratio between the pulsatility index of the middle cerebral artery and the mean pulsatility index value of both uterine arteries.
Oligohydramnios | 24 hours before delivery
  Amniotic fluid index (Assessed acording to four-quadrant technique)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Hernández-Castro, MD PhD, Principal Investigator — Hospital Universitario Dr. José Eleuterio González UANL
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Lebovitz O, Barzilay E, Mazaki-Tovi S, Gat I, Achiron R, Gilboa Y. The clinical value of maternal and fetal Doppler parameters in low-risk postdates pregnancies - a prospective study. J Matern Fetal Neonatal Med. 2018 Nov;31(21):2893-2897. doi: 10.1080/14767058.2017.1359531. Epub 2017 Aug 9. PMID 28738721
- [Background] Lam H, Leung WC, Lee CP, Lao TT. The use of fetal Doppler cerebroplacental blood flow and amniotic fluid volume measurement in the surveillance of postdated pregnancies. Acta Obstet Gynecol Scand. 2005 Sep;84(9):844-8. doi: 10.1111/j.0001-6349.2005.00741.x. PMID 16097973
- [Background] Arabin B, Becker R, Mohnhaupt A, Vollert W, Weitzel HK. Prediction of fetal distress and poor outcome in prolonged pregnancy using Doppler ultrasound and fetal heart rate monitoring combined with stress tests (II). Fetal Diagn Ther. 1994 Jan-Feb;9(1):1-6. doi: 10.1159/000263899. PMID 8142046
- [Background] Tongsong T, Srisomboon J. Amniotic fluid volume as a predictor of fetal distress in postterm pregnancy. Int J Gynaecol Obstet. 1993 Mar;40(3):213-7. doi: 10.1016/0020-7292(93)90833-i. PMID 8096472
- [Background] Adiga P, Kantharaja I, Hebbar S, Rai L, Guruvare S, Mundkur A. Predictive value of middle cerebral artery to uterine artery pulsatility index ratio in hypertensive disorders of pregnancy. Int J Reprod Med. 2015;2015:614747. doi: 10.1155/2015/614747. Epub 2015 Feb 1. PMID 25763408